CLINICAL TRIAL: NCT06742970
Title: Impact of a Telematic Intervention Based on Exercise, Nutrition and Education on Frailty Reversion and Prognosis Among Older Patients with Aortic Stenosis Undergoing Transcatheter Aortic Valve Intervention: the TELE-FRAIL TAVI Clinical Trial
Brief Title: Telematic Intervention for Reversing Frailty Among Older Patients with Aortic Stenosis Undergoing Transcatheter Aortic Valve Intervention. the TELE-FRAIL TAVI Clinical Trial
Acronym: TELEFRAIL TAVI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Blanca Miranda Serrano, Dr, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TELE-FRAIL TAVI
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Aortic Stenosis
Keywords: frailty; aortic stenosis; TAVI; exercise; nutrition; older
MeSH Terms: conditions — Aortic Valve Stenosis; Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care after TAVI (No Intervention): 3 months usual care after TAVI
- Telematic intervention (Experimental): Telematic intervention will be performed by a specialized company hired by the investigational team.
  Trained nurses will contact patients assigned to the intervention groups by videocalls at weeks 1,3,5,7,9,11 and 12 after the admission. The specialized nurses will supervise the exercise program sessions (based on an adaptation of he VIVI FRAIL program), correcting potential mistakes and recommending the optimal way for performing the training program. Patients will take a 200 ml dose of hyperproteic, hypercaloric nutrition supplements daily one hour after performing the exercise session. Information about the optimal diet adapted to the clinical profile of patients will be also provided. Additionally, health information about the disease, the importance of adherence to treatments and recommendations and the best measures for controling cardiovascular risk factors, comorbidities and avoiding clinical complications will be also provided
  Interventions: Combination Product: Telematic intervention

INTERVENTIONS:
Combination Product: Telematic intervention — Telematic intervention will be performed by a specialized company hired by the investigational team. Trained nurses will contact patients assigned to the intervention groups by videocalls at weeks 1,3,5,7,9,11 and 12 after the admission. The specialized nurses will supervise the exercise program sessions (based on an adaptation of he VIVI FRAIL program), correcting potential mistakes and recommending the optimal way for performing the training program. Patients will take a 200 ml dose of hyperproteic, hypercaloric nutrition supplements daily one hour after performing the exercise session. Information about the optimal diet adapted to the clinical profile of patients will be also provided. Additionally, health information about the disease, the importance of adherence to treatments and recommendations and the best measures for controling cardiovascular risk factors, comorbidities and avoiding clinical complications will be also provided
  Arms: Telematic intervention

SUMMARY:
The TELE FRAIL clinical trial is a randomized trial designed to compare, among older frail patients with aortic stenosis undergoing transcatheter valve intervention (TAVI), the impact of usual care after vs a telematic intervention (including a supervised exercise training program, nutrition and education) on frailty reversal and clinical outcomes three months after the TAVI procedure.

The trial will include older patients a with baseline frailty criteria with severe AS undergoing TAVI. A comprehensive geriatric assessment will be performed after the TAVI procedure in all patients.

Inclusion criteria will be: a) patients aged 75 years or older; b) severe symptomatic aortic stenosis, as defined by a mean aortic gradient≥40 mmHg and/or an aortic valve area < 1cm2 measured by transtoracic echocardiography; c) performance of successful TAVI during the admission, and d) baseline frailty criteria, as defined by Short Physical Performance Battery test value <10 and a FRAIL scale value ≥3.

Exclusion criteria will be: a) negative to participate in the trial; b) unability to undergo a comprehensive geriatric assessment or study related procedures ; c) unability to complete clinical follow up, and d) life expectancy lower than one year.

Patients will be randomized (1:1) to intervention or control arms before hospital discharge after the TAVI procedure.

Patients assigned to the intervention will undergo a telematic intervention during the first 90 days after the admission. Trained nurses form an specialized company will contact patients by videocalls at weeks 1,3,5,7,9,11 an12 months. This telematic intervention will include 1) a supervised exercise program (based on an adaptation of the VIVI-FRAIL program) during this 12 weeks; 2) nutrition intervention: The investigator team will provide patients with nutrition supplements for the first 12 weeks after the admission. Patients will take daily a dose of 200 ml of hypercaloric hyperproteic supplements one hour after performing the corresponding exercise training session. Patients will also receive information about the optimal dieta adapted to their clinical profile; and c) health education about the disease, the importance of adherence to medical treatments and recommendations and the best measures for preventing complications.

Main outcome measured will be the proportion of patients with frailty (as measured by a Short Physical Performance Battery test value <10) 3 months after the admission.

Secondary outcomes will include 1) the number of days alive out of hospital during the first year, 2) need for readmission at 3 months and at one year, 3) overall mortality at one year, 4) incidence of cardiovascular events (myocardial infarction, need for unplanned revascularization or stroke) at 3 months and at one year, 5) proportion of frail patients (SPPB<10) at one year, 6)disability for acitivies of daily living (Barthel index) at three months and at one year, 7) nutritional risk (as measured by the MA-Sf test) at three months and at one year and 8) quality of life (as defined by the EQ-5D-5L test) at three months and at one year.

DETAILED DESCRIPTION:
**Introduction** Degenerative aortic stenosis (AS) is the most common valvular disease in Western countries, largely due to increased life expectancy and the progressive aging of the population. Percutaneous aortic valve replacement (TAVI) has revolutionized the treatment of AS, demonstrating its effectiveness in inoperable patients, high-risk patients, and recently even in patients with low or intermediate surgical risk. This increasing evidence has led to a steady rise in TAVI procedures annually, generating a need for healthcare systems to adapt and optimize healthcare pathways and hospital stays.

AS is a disease predominantly associated with aging. The presence of frailty, comorbidities, and other geriatric syndromes is strongly linked to complications, the need for readmissions, and mortality both in conservatively treated patients and those undergoing surgery or TAVI. Frailty and comorbidity burden are also associated with a higher incidence of procedure-related complications, despite technological advances making TAVI increasingly less invasive. Previous data suggest that patients with greater comorbidity burden have higher rates of readmission and extracardiac mortality, which can limit the benefit of TAVI and even negate it in some highly comorbid patients. Therefore, optimizing patient selection to avoid the futility of the procedure remains a key clinical challenge.

Frailty is a phenotype characterized by vulnerability to potential external stressors, and it may be reversible. In patients with cardiovascular diseases, a significant part of frailty is due to heart disease itself, and therefore potentially reversible with its specific treatment. However, in patients with a higher comorbidity burden, it can be challenging to determine what proportion of frailty is due to other health conditions. It has been suggested that managing frail patients requires a comprehensive approach for frailty reversal, including physical exercise, proper nutrition, and strict control of comorbidities that may accelerate frailty progression. Some publications have shown that physical exercise programs can partially reverse frailty in various cardiovascular settings, including AS patients. However, implementing these strategies in clinical practice presents significant challenges, including the cost of enrolling a growing number of patients in cardiac rehabilitation programs and the difficulty in achieving sustained adherence to these programs.

Telemedicine presents potential advantages, especially in managing elderly patients with frailty and cardiovascular diseases, by enabling proper follow-up while avoiding logistical barriers such as transportation and suboptimal adherence, particularly relevant in this context. Different telemedicine-related tools have proven useful in improving outcomes for patients with heart failure by detecting early decompensation and preventing hospital admissions and other complications. However, there is no experience with applying telemedicine to frail patients with AS undergoing TAVI.

The primary objective of the TELE-FRAIL TAVI clinical trial is to analyze the effect of a comprehensive telehealth intervention on frailty reversal at 3 months post-TAVI compared to standard management in patients with AS undergoing TAVI.

**Methods**

**Study Design** This is a prospective, multicenter, randomized (1:1) study designed to compare a comprehensive telehealth intervention for frailty versus usual post-discharge management in patients aged ≥75 years with AS and frailty criteria undergoing TAVI. The study will be conducted across 20 hospitals in Spain, involving clinical and interventional cardiologists, geriatricians, and other experts in managing these patients, as well as trained nursing staff.

**Study Population**

* Inclusion Criteria:** Patients eligible for inclusion are those who meet the following criteria: 1) Severe AS, defined as a mean aortic gradient >40 mmHg or aortic valve area <0.8 cm² on echocardiography; 2) Age ≥75 years; 3) Underwent TAVI during hospitalization; 4) Baseline frailty criteria (pre-procedure) defined as a score of <10 on the Short Physical Performance Battery (SPPB) and a score of ≥3 on the FRAIL scale.
* Exclusion Criteria:** 1) Refusal to participate in the study; 2) Inability to perform geriatric assessments or comply with study procedures; 3) Inability to understand or sign informed consent; 4) Life expectancy <12 months.

In addition to the defined criteria, the inclusion of the patient in the study and the derived procedures must be deemed reasonable by the medical team responsible for the patient. Any complications that arise during hospitalization must be reasonably resolved as a prerequisite for inclusion in the study.

**Treatment Protocol**

Before undergoing the TAVI procedure, a baseline geriatric evaluation will be conducted through an interview with the patient and/or family or caregivers. This evaluation will be multidisciplinary, involving trained staff from the participating centers and will include:

* Functional capacity for basic daily activities, assessed by the Barthel Index.
* Instrumental activities, assessed by the Lawton-Brody Index.
* Cognitive status assessed by the Pfeiffer Test, as well as the Mini Mental State Examination.
* Frailty assessment using the SPPB.
* Comorbidity assessment using the Charlson Index, with a maximum score of 37 points.

Patients with frailty criteria who agree to participate in the study will be randomized before hospital discharge (after TAVI) into two possible treatment arms: a) Comprehensive telehealth intervention (nutrition + supervised physical exercise + health education) for the first 90 days; or b) Usual post-discharge management. Randomization will be computer-generated in a 1:1 ratio.

**Frailty Intervention** The intervention will be carried out telematically in the first 90 days post-discharge by a specialized company. Healthcare professionals specialized in nutritional support and physical exercise adapted to frail patients will conduct weekly video calls after discharge, followed by calls at 15 days and every 2 weeks for the first 3 months. The physical exercise program will use an adaptation of the VIVI FRAIL program.

* Nutritional Support:** Patients assigned to the frailty intervention arm will receive appropriate nutritional information tailored to their profile after hospital discharge. Nutritional supplements will be provided for the first 3 months post-discharge, consisting of a hypercaloric and hyperproteic formula taken once daily after completing the exercise regimen.
* Health Education:** During video calls over the first 3 months, patients will receive additional information on nutrition and exercise, and any questions will be answered. Patients will also be provided with information to optimize adherence to therapeutic regimens and control cardiovascular risk factors.

**Outcome Measures**

The primary outcome measure is the percentage of patients with frailty reversal, measured by SPPB (i.e., achieving an SPPB score ≥10) at 3 months post-discharge. Secondary outcomes include:

* Number of days alive and out of hospital during the first year post-TAVI.
* Readmission rate (cardiac and non-cardiac causes) at 3 months and 1 year post-TAVI.
* Overall and cardiovascular mortality at 3 months and 1 year post-TAVI.
* Incidence of cardiovascular events (myocardial infarction, stroke, or revascularization) at 1 year post-TAVI.
* Percentage of patients remaining robust (SPPB >10) at 1 year post-TAVI.
* Disability (defined by Barthel Index at 3 months and 1 year post-TAVI).
* Nutritional risk (defined by MNA-SF at 3 months and 1 year post-TAVI).
* Quality of life (defined by EQ-5D-5L at 3 months and 1 year post-TAVI).

**Geriatric Evaluation During Follow-Up** This will be conducted in-person by trained personnel at participating centers, blinded to the treatment arm. The following aspects will be reevaluated at 3 months and 1 year: functional capacity (Barthel Index), instrumental activities (Lawton-Brody Index), nutritional risk (MNA-SF), cognitive capacity (Pfeiffer Test), quality of life (EQ-5D-5L), and frailty using FRAIL, Clinical Frailty Scale, SPPB, and Essential Frailty Toolset scales. Clinical follow-up includes an in-person clinical visit at 3 months and 1 year.

**Study Committees** This project is an independent clinical trial with no funding from the industry, promoted by the investigative team. A steering committee will be responsible for supervising the scientific and operational aspects of the study. Patients and investigators will not be blinded to treatment arm allocation, but clinical events will be evaluated by an event adjudication committee blinded to treatment allocation to avoid bias. Similarly, a data safety monitoring board will be responsible for making pertinent recommendations to the steering committee regarding the outcome measures and any possible safety observations.

**Statistical Analysis and Sample Size** Previous data from elderly patients with AS and frailty criteria treated with TAVI show an approximate 50% frailty reversal rate after the TAVI procedure. Assuming an estimated 70% frailty reversal in the telehealth intervention arm, with an 80% statistical power, a bilateral alpha error of 0.05, and assuming a 10% loss to follow-up, a sample size of 206 patients (103 patients per arm) is calculated. To achieve the proposed sample size, a multicenter approach is necessary.

All statistical comparisons will be made under the intention-to-treat principle. Results will be presented as frequencies and percentages or median (standard deviation), as appropriate. Group comparisons will be conducted using Fisher's exact test. Patient follow-up will be censored at the time of death or the end of the study. Primary outcome measures will be compared between the two groups using a logistic regression model, considering frailty reversal as the dependent variable, the intervention as the fixed independent variable, and other covariates with significant association included in the final statistical model. In addition to the secondary outcome measures, the effect of the intervention on clinical events will be described using a Kaplan-Meier method, with a Cox regression model employed for evaluation. Hazard ratios (HR) and their 95% confidence intervals (CI) will be calculated. For all analyses, a p-value <0.05 will be considered statistically significant. Pre-specified subgroup analyses will be performed based on gender and comorbidity burden (Charlson Index).

**Ethical Aspects** Participants and their families will receive detailed information about the risks and potential benefits of study participation. Informed consent documents will be evaluated by the relevant ethics committee. Participants will be given the opportunity to carefully read the consent document and ask questions before signing it. All participants must sign the informed consent document before inclusion in the study. A copy of the consent document will be provided to participants. The rights and welfare of participants will be protected, emphasizing that the quality of medical care will not be negatively affected if they refuse to participate in the study.

**Discussion** Despite TAVI being established as the treatment of choice for the majority of elderly patients with AS, avoiding futility in patients with high comorbidity burden, frailty, and disability remains a clinical challenge. A significant percentage of elderly patients with AS exhibit frailty, partly due to their heart condition (which can be potentially reversed with specific treatment) and partly due to other comorbidities. It has been described that in patients with greater comorbidity burden, treating their AS in isolation may not provide clinical benefit in the absence of other measures. Understanding each patient's profile in detail is crucial for correctly managing AS and their overall condition once valvulopathy has been corrected.

Frailty is considered an intermediate state in the transition to disability that is potentially reversible, especially in its early stages. For this reason, a holistic multidisciplinary approach is important, supported by pillars such as physical exercise, adequate nutrition, and strict control of comorbidities. Some exercise programs have been shown to partially reverse frailty in various cardiovascular settings, including AS patients. However, implementing these strategies in clinical practice presents significant logistical challenges, as well as difficulties in achieving sustained adherence to these programs.

The TELE FRAIL TAVI clinical trial aims to analyze the potential impact of a comprehensive intervention on frailty reversal and prognosis in frail elderly patients undergoing TAVI. It is hoped that the telematic nature of the intervention will enable high adherence to recommendations on physical exercise and nutrition, contributing to frailty reversal alongside correction of AS through TAVI. The study design should allow for a description of the percentage of patients in whom frailty reverses through this combined strategy compared to the TAVI and conventional follow-up strategy, as well as a description of the clinical and geriatric profile of patients in whom this strategy fails and for whom TAVI is likely to be futile. Therefore, the results of the TELE FRAIL TAVI clinical trial are expected to provide valuable insights into the management of frail elderly patients with AS undergoing TAVI, with significant clinical, economic, and social implications for optimizing their management and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* older patients with aortic stenosis undergoing TAVI
* baseline frailty criteria (SPPB <10)

Exclusion Criteria:

* unability to sign informed consent
* unability to complete geriatric assessment
* unability to complete follow up

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
frailty 3 months after the admission | 3 months after the admission
  SPPB value <10

CONTACTS AND LOCATIONS:
Locations (1):
- Calle de Nuestra Señora de Guadalupe, Nº 5 y 7 28028, Madrid (España), Madrid, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided
to be defined

REFERENCES:
- [Derived] Bernal-Labrador E, Romaguera R, Garcia-Blas S, Regueiro A, Serra V, Asmarats L, Tizon-Marcos H, Agudelo V, Scardino C, Casanova-Sandoval JM, Rodriguez-Gabella T, Jimenez-Mendez C, Perez-Rivera A, Robles-Gamboa C, Ayesta A, Diez-Villanueva P, Raposeiras-Roubin S, Amat-Santos IJ, Esteve-Pastor A, Veiga-Fernandez G, Anguita M, Marti-Sanchez D, Martinez-Velilla N, Cortes L, Calvo E, Asimbaya S, Formiga F, Ariza-Sole A. Telematic intervention on frailty in patients undergoing TAVI. Design of the TELE-FRAIL TAVI clinical trial. REC Interv Cardiol. 2025 Jul 10;7(4):223-228. doi: 10.24875/RECICE.M25000519. eCollection 2025. PMID 41333125